CLINICAL TRIAL: NCT02616367
Title: Comparison Between Ropivacaine and Liposomal Bupivacaine Periarticular Injections for Pain Relief After Total Knee Arthroplasty
Brief Title: Comparison of Comparison of Ropivacaine and Liposomal Bupivacaine for Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never initiated
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1503M66201
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Arthroplasty; Replacement; Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liposomal bupivacaine Periarticular injection (Experimental): Will consist of 100 mL (one syringe with 50 mL total: 40 mL 0.25% bupivacaine, 300 mcg epinephrine, 1 mL ketorolac, 2.5 mL morphine, 6.5 mL normal saline) (one syringe with 50 mL total: 20 mL liposomal bupivacaine 30 mL normal saline).
  Interventions: Drug: liposomal bupivacaine Periarticular injection
- Ropivacaine Periarticular Injection (Active Comparator): Will consist of 100 mL (1 mL ketorolac, 2.5 mL morphine, 28.95 mL normal saline, 300 mcg of epinephrine, and 200 mg ropivacaine
  Interventions: Drug: Ropivacaine Periarticular Injection

INTERVENTIONS:
Drug: liposomal bupivacaine Periarticular injection — Liposomal bupivacaine used for a periarticular injection in the knee
  Other Names: Exparel
  Arms: liposomal bupivacaine Periarticular injection
Drug: Ropivacaine Periarticular Injection — Periarticular Injection for the knee with ropivacaine
  Other Names: Norapin
  Arms: Ropivacaine Periarticular Injection

SUMMARY:
This is a randomized prospective outcomes study comparing two groups of patients. One group will receive liposomal bupivacaine for a periarticular injection. The other will receive ropivacaine for periarticular injection for pain relief after Total Knee Arthroplasty. the primary objective of this study is to determine if liposomal bupivacaine provides superior pain control (decreased maximal pain scores within the first 72 hours post surgery) when compared to ropivacaine when injected in a periarticular injection.

DETAILED DESCRIPTION:
The current standard of care at our institution for pain relief in Total Knee Arthroplasty is ropivacaine injectate into the knee for acute postoperative pain relief. This provides pain relief for a duration of 6-18 hours after surgery. All patients in this study will also receive multimodal analgesia following surgery in both arms of the study. This will be the first study to prospectively analyze these two regimens.

Study group 1 (ropivacaine arm) consist of 100 mL (1 mL ketorolac, 2.5 mL morphine, 28.95 mL normal saline, 300 mcg of epinephrine, and 200 mg ropivacaine) Study group 2 will consist of 100 mL (one syringe with 50 mL total: 40 mL 0.25% bupivacaine, 300 mcg epinephrine, 1 mL ketorolac, 2.5 mL morphine, 6.5 mL normal saline) (one syringe with 50 mL total: 20 mL liposomal bupivacaine 30 mL normal saline). The periarticular injection will occur at the end of the procedure. Adequate analgesia will be defined as < 3 VAS at rest and if VAS is greater that 3 adjustments in oral or intravenous pain medications. Postoperatively the study team will evaluate for any signs of complications. Pain scores and opioid usage will be recorded daily while the subject is in the hospital. A quality of recovery survey will be completed at 72 hours post injection. All subjects will be contacted by phone at day 14 to determine if there have been any adverse events and report their pain level.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary total knee arthroplasty surgery 18-80.

Exclusion Criteria:

* Patient on chronic anticoagulation
* Allergy to local anesthetics, nsaids, or opioids
* Patients who remain intubated for one week after surgery or who are unable to provide information as to their feelings of pain post-operatively for the first week post- operatively
* Daily use of opioid for more than three weeks
* Lack of patient cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
pain control measure on pain scale of 1-10 | 72 hours
  to determine if liposomal bupivacaine provides superior pain control (decreased maximal pain control (decreased maximal pain scores) when compared to ropivacaine when injected in a periarticular injection.

SECONDARY OUTCOMES:
decreased maximal pain on pain scale of 1-10 | 72 hours
  Liposomal bupivacaine via a periarticular injection will result in a decreased maximal pain and improved quality of recovery when compared to ropivacaine when injected in a periarticular injection

CONTACTS AND LOCATIONS:
Overall Officials: Roberto D Blanco, Principal Investigator — University of Minnesota